CLINICAL TRIAL: NCT04695483
Title: Reduction of Progesterone Elevation at Trigger in Poor Responder Bologna' Criteria Patients After Controlled Ovarian Stimulation With Long Acting Standard Stimulation Protocol Compared With Conventional Daily Protocol: a Single Center Prospective Randomized Fase IV Trial
Brief Title: Reduction of Progesterone Elevation at Trigger in POR After Long Acting COS Compared With Daily COS: a Prospective Randomized Trial
Acronym: PE-PMA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Enrico Papaleo, MD, IRCCS San Raffaele
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PE-PMA; 2020-004329-21 (EudraCT Number)
Record Dates: First submitted 2020-12-01; First posted 2021-01-05 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility | interventions — follicle stimulating hormone, human, with HCG C-terminal peptide; follitropin beta

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Corifollitropin alpha group (Experimental): Patients treated with Corifollitropin-alpha in a long-acting controlled ovarian stimulation
  Interventions: Drug: Corifollitropin alfa; Drug: Follitropin Beta
- FSH group (Active Comparator): Patients treated with Follitropin beta in a daily controlled ovarian stimulation protocol
  Interventions: Drug: Follitropin Beta

INTERVENTIONS:
Drug: Corifollitropin alfa — Controlled ovarian stimulation long-acting protocol
  Arms: Corifollitropin alpha group
Drug: Follitropin Beta — Daily controlled ovarian stimulation protocol

SUMMARY:
The overarching objective of this research is to generate clinical evidence to argue the benefits of long acting stimulation protocol compared to the daily stimulation protocol in poor ovarian responder bologna' criteria patients after controlled ovarian stimulation. Reduction in the proportion of subjects with progesterone > 1.1 ng/ml on the day of triggering (day + 13) in the experimental group compared to the control group is expected.

DETAILED DESCRIPTION:
Each patient will receive a first visit for infertility where will be collected subject history and baseline information, and meet all the inclusion / exclusion criteria. Eligible patients who agreed to participate will be randomized to either long acting standard COS with corifollitropin alpha or standard COS with daily FSH in a fixed GnRH antagonist protocol. All patients will be allowed to participate in the study only once and a written informed consent will be obtained from all, following consultation and before the initiation of the treatment.

The endocrine profile of all the patients will be evaluated by analysis of serum progesterone, 17b-estradiol (E2), FSH and LH at different time points: basal condition, during stimulation, at the hCG day and at pick-up.

Transvaginal follicular aspiration will be performed by ultrasound guidance 36 hours after hCG administration. The day of pick up oocytes will be fertilized with partner's semen; after 3-5 days, on the base of its evolution, embryo will be transferred. 14 days after embryo-transfer a preg-nancy test will be performed. Follow up in case of obtained pregnancy will be done until 20 weeks of gestation and considered as ongoing pregnancy.

The entire duration of the study is 24 months, the follow up of the last patients enrolled will be 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Indication to IVF treatment
* Normal BMI (18.5-24.9 kg/m2)
* AMH level < 1.1 ng/ml and/or AFC < 5 follicles and/or < 3 oo-cytes retrieved in previous cycle
* Regular menstrual cycles
* Signed informed consent

Exclusion Criteria:

* Freeze all cycles for abnormal bleeding
* PCOS
* History of untreated autoimmune
* Endocrine or metabolic disorders
* Ovarian cystectomy or oophorectomy
* FSH ≥ 20 lU/L

Ages: 25 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 110 (Actual)
Dates: Start 2022-02-22 (Actual); Primary Completion 2024-01-19 (Actual); Study Completion 2024-05-06 (Actual)

PRIMARY OUTCOMES:
Premature progesterone elevation | day 12
  Progesterone > or equal to 1.1 ng/mL at day of trigger

SECONDARY OUTCOMES:
Percentage of freeze-all cycles due to premature progesterone elevation | day 12
Number of oocytes collected at ovum retrieval | day 14
Fertilization rate | day 15
  Percentage of oocytes fertilized
Number of embryos available | Day 17
Pregnancy rate | day 30
  Beta-HCG positive
Ongoing pregnancy | Up to 20 weeks
  Vital fetus at 20 weeks of gestation

CONTACTS AND LOCATIONS:
Overall Officials: Enrico Papaleo, MD, Principal Investigator — IRCCS San Raffaele
Locations (1):
- Enrico Papaleo, Milan, Italy